CLINICAL TRIAL: NCT03654703
Title: Improved Post-Transplant Cyclophosphamide Regimens for Unmanipulated Haploidentical Transplant in Pediatric Patients With Refractory Acute Myeloid Leukemia
Brief Title: Improved Post-Transplant Cyclophosphamide Regimens for Pediatric Patients With Refractory AML
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Capital Research Institute of Pediatrics (Other Government)
Responsible Party: Principal Investigator, Yan Yue, MD,PhD, Capital Research Institute of Pediatrics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIP-2015-AML
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Hematopoietic System--Cancer
Keywords: HSCT, AML， R-AML
MeSH Terms: interventions — Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclophophamide (Experimental): Cyclophosphamide 50mg/kg/day on day+3，+4 after HSCT. Intervention: drugs:Cyclophosphamide.
  Interventions: Drug: Cyclophosphamide
- Placebo (Experimental): 5% GLS（Placebo) 50ml/day on day+3，+4 after HSCT. Intervention: drugs: Placebo other name: placebo (for Cyclophosphamide) 5%Glugose in water 50ml or normal saline
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — cyclophophamide
  Other Names: Cy

SUMMARY:
No more datas about post-transplant cyclophosphamide (PT/Cy) used in pediatric refractory acute myeloid leukemia (R-AML）patients. Investigators reasoned that this group of patients if they have been treated with ablative conditioning regimens for HSCT combined with PT/Cy, under the rapid of immune reconstitution will have better outcomes.

DETAILED DESCRIPTION:
Haploidentical stem cell transplantation (HSCT) is a potentially curative therapy for patients with high risk or refractory acute myeloid leukemia (R-AML). Graft-versus-host disease （GVHD）is a major barrier to achieve success for patients with HSCT. High dose cyclophosphamide given after HLA-matched related and unrelated allogeneic stem cell transplantation for patients with hematologic malignancies is effective single agent (GVHD) prophylaxis in adults and in pediatric benign patients. Data describing outcomes for pediatric maligant patients has not been reported. Investigators have recruited 26 pediatric patients (3 years < age <18 years) between March 2015 to July 2018 with primary induction R-AML treated in investigators' institution for R-AML with modified myeloablative regimen, post-transplant cyclophosphamide (PTCy) has been used as GVHD prophylaxis.

Conditioning regimen of the group of patient consisted Idrabine(IDA,10mg/m2/day) which was administered intravenously for 2 days, from days -14 to -13, total body irritation (TBI, 9 Gy) which was divided into 3 fractions and 3 days from -12 to -10, thymoglobulin (2.5mg/kg/day) was administered for 3 days, from -9 to -7, etoposide (VP-16, 300mg/m2) which was infused intravenously on day -6, cladribine (10mg/m2/day) which was administered for 3 days from -5 to -2 .

ELIGIBILITY:
Inclusion Criteria:

-refractory AML

Exclusion Criteria:

- complete remission AML

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Disease status | 1 year
  Disease status can be measured by test the of (minimal residual disease) MRD via flow cytometry one time each month until one year after HSCT. MRD<0.0001 （complete remission), if not, relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Y Qin, MD, Study Director — Hematology and oncology
Locations (1):
- Yan Yue, Beijing, Chaoyang District, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sugita J, Kagaya Y, Miyamoto T, Shibasaki Y, Nagafuji K, Ota S, Furukawa T, Nara M, Akashi K, Taniguchi S, Harada M, Matsuo K, Teshima T; Japan Study Group for Cell Therapy and Transplantation (JSCT). Myeloablative and reduced-intensity conditioning in HLA-haploidentical peripheral blood stem cell transplantation using post-transplant cyclophosphamide. Bone Marrow Transplant. 2019 Mar;54(3):432-441. doi: 10.1038/s41409-018-0279-1. Epub 2018 Aug 7. PMID 30087460
- [Result] Marani C, Raiola AM, Morbelli S, Dominietto A, Ferrarazzo G, Avenoso D, Giannoni L, Varaldo R, Gualandi F, Grazia D, Lamparelli T, Bregante S, Van Lint MT, Ibatici A, Bovis F, Lemoli RM, Gobbi M, Bacigalupo A, Angelucci E. Haploidentical Transplants with Post-Transplant Cyclophosphamide for Relapsed or Refractory Hodgkin Lymphoma: The Role of Comorbidity Index and Pretransplant Positron Emission Tomography. Biol Blood Marrow Transplant. 2018 Dec;24(12):2501-2508. doi: 10.1016/j.bbmt.2018.07.025. Epub 2018 Jul 21. PMID 30041010
- [Result] Law AD, Salas MQ, Lam W, Michelis FV, Thyagu S, Kim DDH, Lipton JH, Kumar R, Messner H, Viswabandya A. Reduced-Intensity Conditioning and Dual T Lymphocyte Suppression with Antithymocyte Globulin and Post-Transplant Cyclophosphamide as Graft-versus-Host Disease Prophylaxis in Haploidentical Hematopoietic Stem Cell Transplants for Hematological Malignancies. Biol Blood Marrow Transplant. 2018 Nov;24(11):2259-2264. doi: 10.1016/j.bbmt.2018.07.008. Epub 2018 Aug 7. PMID 30009980